CLINICAL TRIAL: NCT05765630
Title: Evaluation of Two New Innovative Haemostasis Tests: Measurement of the Active Form of GTP-bound Rap1b (aRap1b) in Platelets and the Pro and Antithrombotic Balance of Circulating Endothelial Microvesicles (patEMV) (INNOV-CKD Test)
Acronym: INNOV-CKD test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM20_0328; 2020-A01264-35_ (Other: IDRCB)
Record Dates: First submitted 2023-02-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy patients (Active Comparator)
  Interventions: Biological: BLOOD SAMPLES
- CKD patients not receiving antiplatelet agents (Experimental)
  Interventions: Biological: BLOOD SAMPLES
- CKD patients receiving antiplatelet agents (Experimental)
  Interventions: Biological: BLOOD SAMPLES
- Patients with constitutional thrombopathy with RAP1B activation defect (Experimental)
  Interventions: Biological: BLOOD SAMPLES
- Patients with ACS in the previous month treated with antiplatelet agents (Experimental)
  Interventions: Biological: BLOOD SAMPLES

INTERVENTIONS:
Biological: BLOOD SAMPLES — BLOOD SAMPLES

SUMMARY:
The aim of this PROJECT is to develop two biomarkers to assess the thrombotic and hemorrhagic risk of patients with chronic renal failure (CKD) treated with antiplatelet drugs following the occurrence of an acute coronary syndrome (ACS). These biomarkers will help to adapt antiplatelet therapy on an individual basis (intensity, duration of antiplatelet treatment) and thus reduce the risk of thrombotic and hemorrhagic events in this particularly fragile population. The methods for measuring these two highly innovative biomarkers are currently being developed. The first biomarker corresponds to the measurement of an intraplatelet molecule, Rap1b in its active form (aRap1b). The second biomarker is the measurement of the pro-antithrombotic balance of circulating endothelial microvesicles (patEMV), a reflection of endothelial dysfunction. An automated method for biomarker measurement will be developed in partnership with the industrial partners Stago and BioCytex during the project.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (group 1): DFG>70 ml/mn/1.73m2 in CKD-EPi, Age 18-85 years old, Consent required, Affiliated to social security.
* Antiplatelet agents-naïve CKD patients (group 2): DFG<30 ml/mn/1.73m2 in CKD-EPi, Age 18-85 years old, Consent required, Affiliated to social security.
* CKD patients receiving antiplatelet agents (group 3): DFG<30 ml/mn/1.73m2 in CKD-EPi, receiving antiplatelet agents, Age 18-85 years old, consent required, Affiliated with social security.
* Patients with constitutional platelet dysfunction (group 4): DFG>70 ml/min/1.73m2 in CKD-EPi, Age 18-85 years old, Consent required, Social Security Affiliated, Constitutional haemorrhagic syndrome
* Coronary patients (group 5): DFG>70 ml/mn/1.73m2 in CKD-EPi, Age 18-85 years old, Consent required, Social Security Affiliated, Acute Coronary Syndrome in the previous month requiring AAP.

Exclusion Criteria:

* For all the groups : subjects refusing to participate in the study, pregnant or breastfeeding women, minors (except for special consent), adults subject to a legal protection measure or unable to express their consent (persons under guardianship or curatorship), persons deprived of their rights of liberty by judicial or administrative decision (persons in a situation of social fragility), persons at the end of life.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
aRap1b assay reproducibility | 1 year
  intraclass correlation coefficient and its 95% confidence interval (CI) for assessing the reproducibility over time of aRap1b-GTP for subjects from groups 1, 2, 3, and 5.

SECONDARY OUTCOMES:
Reproducibility of pat EMV | 1 year
  intraclass correlation coefficient and its 95% confidence interval (CI) for assessing the reproducibility over time of microvesicle derived functional assays for subjects from groups 1, 2, 3, and 5.
Repeatability | 1 year
  Coefficient of variation will be determined for different levels of concentration of the analytes (aRap1b resting and activates states and pat EMV)
Analytical specificity | 1 year
  Best threshold values between samples containing the analyte (aRap1B) compared to negative samples which do not contain the analyte.
Range of values in each group | 1 year
  Mean, standard deviation, median, interquartile range

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BONELLO, Pr., Principal Investigator — Service cardiologie Hopital Nord
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France